CLINICAL TRIAL: NCT06807580
Title: Effects of Oral Progesterone in Transgender Women on Breast Development, Sleep Quality, Psychological Distress, and Cardiovascular Risk
Brief Title: Progesterone in Gender Affirming Hormone Therapy Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00006161; 2025P011358 (Other: Emory IRB)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Transgender Women
Keywords: Gender affirming hormone therapy; Transgender women; Progesterone
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Group A will serve as our control group with participants on their existing gender-affirming therapy in addition to a placebo pill.
  Laboratory assessments including estradiol, lipid profile, and Complete metabolic profile (CMP) will be performed at screening.
  Interventions: Drug: Placebo
- Group B (Experimental): Group B will serve as our intervention group with participants on their existing gender-affirming therapy in combination with 200 mg oral micronized progesterone at bedtime.
  Laboratory assessments including estradiol, lipid profile, and Complete metabolic profile (CMP) will be performed at screening.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Placebo — The placebo will be nearly identical in size, color, and shape to micronized progesterone
  Arms: Group A
Drug: Progesterone — Oral micronized progesterone 200 mg
  Other Names: Prometrium 200mg
  Arms: Group B

SUMMARY:
This study aims to study the effects of Oral Progesterone in Transgender Women. The primary goal is to study the effect of progesterone on psychological distress and secondarily on sleep quality, breast size, quality of life and gender congruence and cardiovascular risk.

DETAILED DESCRIPTION:
The transgender population in the U.S. has grown significantly, highlighting a lack of comprehensive research on the safety and efficacy of gender-affirming hormone therapy (GAHT). For transgender females, GAHT typically includes estrogen and an anti-androgen. Recently, there has been growing interest in adding progesterone, based on anecdotal reports of improved breast development and quality of life. However, progesterone's role in transgender women remains unclear.

Studies have linked progesterone (mainly cyproterone acetate) to increased risks of meningiomas, elevated prolactin levels, decreased testosterone, reduced HDL levels, and higher venous thromboembolism (VTE) risk. Cyproterone acetate, often studied in these contexts, is not FDA-approved in the U.S. due to hepatotoxicity, and its use in GAHT is rare. Limited research exists on micronized progesterone, the form most commonly prescribed.

A recent study on low-dose micronized progesterone found no significant effects on sleep quality, psychological distress, or breast development. To address research gaps, a new study aims to evaluate higher-dose micronized progesterone's impact on cardiovascular risk, sleep quality, breast development, and psychological distress over a longer period. The hypothesis suggests neutral effects on breast development, sleep, and quality of life, with potential negative to neutral cardiovascular effects.

Given the lack of recommendations for or against progesterone in GAHT, further research is critically needed.

ELIGIBILITY:
Inclusion Criteria:

- Participants will be transgender women, who have been on gender-affirming hormone therapy for at least 6 months before the start of the study.

Exclusion Criteria:

* Peanut allergy
* Liver disease (liver enzyme elevations and/or evidence of acute or chronic hepatitis). In our lab, the upper limit of normal for aspartate aminotransferase (AST) is 39, and the upper limit of normal for alanine aminotransferase (ALT) is 52.
* Stage 4/5 chronic kidney disease
* Congestive heart failure
* Medical disease or medication use associated with gynecomastia (i.e tumor, hyperthyroidism, chronic kidney disease, cirrhosis, ACE inhibitors, statins, haloperidol, tricyclic antidepressants, atypical antipsychotics)
* Pre-existing cardiovascular disease
* Prior or current history of thromboembolism, known clotting disorders, current or recent anti-thrombotic therapy for venous thromboembolism.
* History of breast cancer
* Prior progesterone use
* Uncontrolled depression and/or suicidal ideation
* Current hypothyroidism (even if controlled with treatment) Progesterone in Gender Affirming Hormone Therapy 9 Version #4, 10/30/24
* Cannabis use of greater than 1 use/week in the past 3 months
* Previously identified BRCA 1 or 2 gene mutation or other familial breast cancer.
* Abnormal mammogram (if indicated - for patients above the age of 50 and on estrogen for 5 or more years OR positive family history of breast cancer) with results of BIRADS 3 or higher. Subjects with a BIRADS 0 mammogram must have undergone additional imaging demonstrating BIRADS 1 or 2 prior to enrollment.
* Have had or are planning to undergo breast enhancement or gender affirming top surgery in the next 6 months
* Uncontrolled hypertension, defined as systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mmHg.
* Triglycerides ≥ 500 mg/dL.
* In our lab, the upper limit of normal for aspartate aminotransferase (AST) is 39, and the upper limit of normal for alanine aminotransferase (ALT) is 52.
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2.
* Estradiol levels outside the stable range (100-300 pg/mL)
* Heavy smoking, defined as 25+ cigarettes per day
* Non-English speaking or those with limited English proficiency

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants will be transgender women
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | Baseline, Month 6
  Kessler Psychological Distress Scale (K10) scale will be used to measure distress.
  This is a 10-item questionnaire intended to yield a global measure of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4 week period.
  The numbers attached to the patients 10 responses are added up and the total score is the score on the Kessler Psychological Distress Scale (K10). Scores will range from 10 to 50. People seen in primary care who:
  * score under 20 are likely to be well
  * score 20-24 are likely to have a mild mental disorder
  * score 25-29 are likely to have moderate mental disorder
  * score 30 and over are likely to have a severe mental disorder

SECONDARY OUTCOMES:
Effect of progesterone on breast development | Baseline, Month 6
  Breast size will be measured using hemi-circumference. Hemi circumference will be measured as the medial breast infliction point, the most medial point of the breast across the nipple level to the lateral breast inflection point.
Effect of progesterone on sleep quality | Baseline, Month 6
  Sleep quality will be measured by having participants from both Group A and B take the 19 item Pittsburgh sleep index. The Pittsburgh Sleep Quality Index (PSQI) is a 19-item questionnaire that assesses sleep quality and disturbances over the past month.
  Each item is scored on a scale of 0-3, with 3 being the worst. The global score ranges from 0-21, with higher scores indicating worse sleep quality.
Effect of progesterone on gender congruence | Baseline, Month 6
  The gender Congruence and Life Satisfaction Scale (GCLS) will be used. It is a 38-item scale with each item scored on a 5-point scale.
  Items are scored on a 5-point scale (always = 1; never = 5). A higher score indicates a more positive outcome (higher gender congruence, better gender-related mental well-being, and better general life satisfaction).
Effect of progesterone on cardiovascular risk | Baseline, Month 6
  Change in lipid profile from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Transgender Clinic, Atlanta, Georgia, United States